CLINICAL TRIAL: NCT06408519
Title: Open -Label Placebo for Non-specific Pain in the Emergency Department: Study Protocol for a Mixed-method Randomised Control Feasibility Study
Brief Title: Open-Label Placebo for Non-Specific Pain in the ED
Acronym: OLP_EM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruno Minotti (Other)
Collaborators: Roland Bingisser, Principal Investigator, Head of Emergency Department, University Hospital Basel (Unknown); Jens Gaab, Co-investigator, Head of Division University of Basel, Faculty of Psychology (Unknown); Bojana Degen, Co-investigator, University of Basel, Faculty of Psychology (Unknown); Anna Szczesna, Co-investigator, University Hospital Basel, Emergency Department (Unknown); Christian H Nickel, Co-investigator, Deputy Head of Emergency Department, University Hospital Basel (Unknown)
Responsible Party: Sponsor-Investigator, Bruno Minotti, Sponsor Investigator, University Hospital Basel, Emergency Department, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-00089; am24Bingisser
Record Dates: First submitted 2024-04-25; First posted 2024-05-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pain, Acute
Keywords: open-label placebo; non-specific pain; emergency department
MeSH Terms: conditions — Acute Pain; Emergencies | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: mixed-method randomised control feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-label Placebo (Experimental): Treatment with open-label placebo pills 3x/day
  Interventions: Other: Placebo (open-label)
- Treatment as usual (Active Comparator): Treatment as usual defined as Ibuprofen 3x/day
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Other: Placebo (open-label) — P-Tabletten weiss 10mm (Lichtenstein, Zentiva) pills 3x/day
  Arms: Open-label Placebo
Drug: Ibuprofen 400 mg — Ibuprofen pills 3x/day
  Other Names: Ibuprofen-Sandoz
  Arms: Treatment as usual

SUMMARY:
The aim of this study is to assess whether an intervention with open-label placebo (OLP) for non-specific pain in the emergency department is feasible.

DETAILED DESCRIPTION:
This project is a collaboration between the Emergency Department at the University Hospital of Basel and the Faculty of Psychology at the University of Basel. The investigation will analyze whether an intervention consisting of open-label placebo tablets is feasible for patients with non-specific pain in the emergency department. Open-label placebos are administered without deception, meaning the patients are aware they are taking a placebo. Patients will be randomized into intervention group (OLP) or control group (treatment as usual) with ibuprofen. The study duration for patients is 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of non-specific acute pain
* Able to understand the study and its outcome measures
* Signed informed consent
* 18 years or older
* Sufficient German language skills

Exclusion Criteria:

* Chronic pain
* Treatment with pain medication for > 7 days prior to ED visit
* Known allergy or intolerance to ibuprofen
* Known hereditary galactose-intolerance, lactase deficiency or glucosegalactose malabsorption
* Participation in another clinical trial with medicinal products
* Need for hospitalization
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of eligible patients consenting to participate | 12 months
  Feasibility Outcome. Threshold: ≥30% of eligible patients for the target population of 50 patients within 12 months.
Rate of patients adhering to the study protocol in terms of medication intake | 7 days
  Feasibility Outcome. Threshold: ≥70% of patients with at least ≥70% medication intake according to the protocol.
Rate of patients completing their outcome (self-)assessments (i.e. questionnaires) | 30 days
  Feasibility Outcome. Threshold: ≥80% of patients with completed assessments/questionnaires..
Rate of patients' satisfaction with the intervention and study procedure | 30 days
  Feasibility Outcome. Threshold: ≥70% of patients with a score ≥6 on a scale from 0 (absolutely not satisfied) to 10 (absolutely satisfied).

SECONDARY OUTCOMES:
Change in pain intensity as measured through daily self-reported Brief Pain Inventory-Short Form (BPI-SF) | 8 days
  Clinical Outcome (exploratory). Score from 0 (no pain) to 10 (worste pain ever) for each pain severity subscale of the BPI-SF (minimal, average, and maximal pain intensity in the last 24 hours).
Change in pain interference as measured through daily self-reported Brief Pain Inventory-Short Form (BPI-SF) | 8 days
  Clinical Outcome (exploratory). Score from 0 (no impact of pain) to 10 (maximal impact of pain) for each pain interference subscale of the BPI-SF (impact of pain in the last 24 hours on mood, sleep, activity, work, social relationships, enjoyment of life).
Use of rescue medication | 8 days
  Clinical Outcome (exploratory). Proportion of patients requiring rescue medication (including amount of rescue medication intake) in both arms during the first 8 days.
Frequency and nature of side effects, adverse events | 30 days
  Clinical Outcome (exploratory)
Rate of patients with ED re-attendance | 30 days
  Clinical Outcome (exploratory)
Average pain intensity 30 days after the ED index visit | 30 days
  Clinical Outcome (exploratory). Measured with a score from 0 (no pain) to 10 (worste pain ever) for each pain severity subscale of the BPI-SF (minimal, average, and maximal pain in the last 24 hours).
Average pain interference 30 days after the ED index visit | 30 days
  Clinical Outcome (exploratory). Measured with a score from 0 (no impact) to 10 (maximal impact) for each pain interference subscale of the BPI-SF (impact of pain in the last 24 hours on mood, sleep, activity, work, social relationships, enjoyment of life).
Frequency of medication use between day 8 and 30 | 30 days
  Clinical Outcome (exploratory). Frequency of (optional) medication use between day 8 and 30.
Rate of patients with specific cause of pain within 30 days of the index visit | 30 days
  Clinical Outcome (exploratory). Rate and type of diagnosis of a specific cause of pain following the index visit (i.e. in the course, e.g. appendicitis diagnosed after presenting with "non-specific abdominal pain" at the index visit).
Depression measured by depression scale of the German version of the Patient Health Questionnaire (PHQ-9) at different timepoints. | 30 days
  Clinical Outcome (exploratory). PHQ-9 score from 0 (no depression) to 27 (severe depression).

OTHER OUTCOMES:
Rate of eligible patients declining consent | 1 day
  Additional variables of interests. If communicated (NOTE: not mandatory according to Good Clinical Practice), the reason for declining will also be recorded for anonymous qualitative analysis.
Expectancy of Pain Relief Scale on the day of index visit | 1 day
  Additional variables of interests. Score from 0 (no expectancy of pain relief) to 10 (maximum expectancy of pain relief).
Desire for Pain Relief Scale on the day of index visit | 1 day
  Additional variables of interests. Score from 0 (no desire of pain relief) to 10 (maximum desire of pain relief).
Placebo understanding during day of index visit | 1 day
  Additional variables of interests. Qualitative analysis (open questions) on placebo understanding.
Placebo beliefs during day of index visit | 1 day
  Additional variables of interests. Qualitative analysis (open questions) on placebo beliefs.
Placebo intervention credibility during the index visit | 1 day
  Additional variables of interests. Qualitative analysis (open questions) on placebo credibility.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Minotti, MD, Study Chair — Emergency Department, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Degen B, Szczesna A, Nickel CH, Bingisser R, Gaab J, Minotti B. Open-label placebo for non-specific pain in the emergency department (OLP EM): study protocol for a mixed-method randomised control feasibility study in Switzerland. BMJ Open. 2025 Mar 25;15(3):e090508. doi: 10.1136/bmjopen-2024-090508. PMID 40132833